CLINICAL TRIAL: NCT03433183
Title: SARC031: A Phase 2 Trial of the MEK Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate) in Combination With the mTOR Inhibitor Sirolimus for Patients With Unresectable or Metastatic Malignant Peripheral Nerve Sheath Tumors
Brief Title: SARC031: MEK Inhibitor Selumetinib (AZD6244) in Combination With the mTOR Inhibitor Sirolimus for Patients With Malignant Peripheral Nerve Sheath Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC031; CDMRP-NF150092 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-01-29; First posted 2018-02-14 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-03

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors; Neurofibromatosis 1
MeSH Terms: conditions — Neurofibrosarcoma; Neurofibromatosis 1 | interventions — AZD 6244; Sirolimus

STUDY DESIGN:
Intervention Model Description: A Simon's two-stage phase 2 trial of MEK inhibitor selumetinib in combination with the mTOR inhibitor sirolimus to determine the safety and clinical benefit in patients with unresectable or metastatic MPNST
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selumetinib and Sirolimus (Experimental): A Simon's two-stage phase 2 trial of MEK inhibitor selumetinib in combination with the mTOR inhibitor sirolimus to determine the safety and clinical benefit in patients with unresectable or metastatic MPNSTs. Both agents will be given orally on an empty stomach. Selumetinib will be given orally at a dose of 50mg twice daily continuously. Sirolimus will be given orally at a dose of 4mg once daily with a cycle 1 day 1 loading dose of 12mg. Each cycle will be considered 28 days.
  Interventions: Drug: Selumetinib; Drug: Sirolimus

INTERVENTIONS:
Drug: Selumetinib — Selumetinib (AZD6244) is an oral selective inhibitor of the mitogen-activated protein kinase (MEK) 1/2 currently in development for adult malignancies, pediatric low-grade gliomas and NF1 plexiform neurofibromas. MEK is a critical kinase in the mitogen activated protein (MAP) kinase signal transduction pathway for many growth factor receptors that provide growth signals to cancer cells.
  Other Names: AZD6244
Drug: Sirolimus — Sirolimus is a macrocyclic lactone produced by Streptomyces hygroscopicus and inhibitor of mammalian Target of Rapamycin (mTOR) serine threonine kinase, which plays a critical role in regulating cellular energy sensing, growth and metabolism.
  Other Names: Rapamycin

SUMMARY:
To determine the clinical benefit rate of selumetinib in combination with sirolimus in patients with unresectable or metastatic neurofibromatosis type 1 (NF1) associated or sporadic MPNST.

DETAILED DESCRIPTION:
I. Primary Objective

• To determine the clinical benefit rate of selumetinib in combination with sirolimus in patients with unresectable or metastatic NF1 associated or sporadic MPNST

II. Secondary Objective(s)

* To define and describe the toxicities of selumetinib in combination with sirolimus in patients with unresectable or metastatic NF1 associated or sporadic MPNST.
* To assess the impact on intensity and pain interference and correlate to changes in clinical, imaging response and progression
* To assess progression free and overall survival

Selumetinib will be given orally 50mg twice daily continuously and sirolimus will be given orally 4mg once daily with a cycle 1 day 1 loading dose of 12mg. One cycle will be 28 days. Patients will be able to remain on treatment as long as they do not experience progressive disease or unacceptable toxicity. Stage 1 will require 7 patients, with no further accrual if 0 of 7 respond. If 1 or greater of the 7 patients respond, accrual will continue until 21 patients have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years of age
* Patients with unresectable or metastatic histologically confirmed sporadic or NF1 associated MPNST.
* Patients must have measureable disease by RECIST.
* Patients must have experienced progression after one or more prior regimens of cytotoxic chemotherapy. Patients who have refused cytotoxic chemotherapy or for whom treatment on this protocol prior to receiving cytotoxic chemotherapy is felt to be in the best interest for the patient by the local investigator will also be eligible.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering on this study.
* No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study entry.
* The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry.
* The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.
* The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry.
* The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.
* At least 2 months post-autologous stem cell transplant or at least 3 months post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease and on stable doses of immunosuppressive medications if required.
* The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.
* No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) is permitted.
* Karnofsky performance level ≥ 50%.
* Patients who are unable to walk because of paralysis or motor weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
* Peripheral absolute neutrophil count (ANC) of ≥1000/μL
* Platelet count ≥75,000/μL (transfusion independent (no transfusion within at least 7 days prior to enrollment)
* Total bilirubin must be ≤ 1.5 times the upper limit of normal (ULN)
* SGPT (ALT) must be ≤ 3.0 times ULN
* Serum creatinine ≤ ULN or creatinine clearance >60 ml/min/1.73 m2
* Serum triglyceride level ≤300 mg/dL and serum cholesterol level ≤ 300 mg/dL (Patient may be on lipid-lowering medicine)
* Normal ejection fraction by ECHO or cardiac MRI >55%
* QTcF ≤ 450ms
* Fertile men and women of childbearing potential must agree to use an effective method of birth control.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of clinical progression or stable disease at 4 weeks.

Exclusion Criteria:

* Patients receiving other anti-cancer agents are not eligible.
* Patients who cannot swallow whole pills.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent (for example cyclosporine). Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunizations with attenuated live vaccines within four weeks of study entry or during study period.
* Any recent major surgery within a minimum of 4 weeks, with the exception of surgical placement for vascular access, or minor surgery (excluding tumor biopsies) within 14 days.
* Patients who any known severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Severely impaired lung function defined as spirometry and DLCO that is 50% of the normal predicted value corrected for hemoglobin and alveolar volume and/or O2 saturation that is 88% or less at rest on room air. For patients who do NOT have respiratory symptoms (e.g. dyspnea at rest, known requirement for supplemental oxygen), pulmonary function test is not required.
  * Cardiac conditions as follows:

    * Uncontrolled hypertension (blood pressure ≥150/95 mmHg despite medical therapy).
    * Acute coronary syndrome within 6 months prior to starting treatment
    * Uncontrolled angina despite medical therapy
    * Symptomatic heart failure NYHA Class II-IV prior or current cardiomyopathy, or severe valvular disease
    * Prior or current cardiomyopathy
  * Uncontrolled Type 1 or 2 diabetes as defined by fasting serum glucose >1.5 x ULN
  * Uncontrolled infection
  * Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome, or renal tubular acidosis.
  * Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of small bowel, symptomatic inflammatory bowel disease, or ulcerative colitis, or partial or complete bowel obstruction.
  * Ophthalmological conditions as follows:

    * Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion
    * Intraocular pressure (IOP) > 21 mmHg or uncontrolled glaucoma
* Supplementation with vitamin E greater than 100% of the daily recommended dose.
* Hypersensitivity to active or inactive excipients of rapamycins (sirolimus, temsirolimus or everolimus) or selumetinib or drugs with similar chemical structures or class to sirolimus or selumetinib.
* Patients unwilling or unable to comply with the protocol.
* Seville orange, star fruit, grapefruit and their juices, and St. John's Wort use are not allowed while on study.
* Exposure to strong or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP if taken within the stated washout periods before the first dose of study treatment.
* Exposure to specific substrates of drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K within the appropriate washout periods (a minimum of 5 x reported elimination half-life) before the first dose of study treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate of selumetinib in combination with sirolimus in patients with unresectable or metastatic NF1 associated or sporadic MPNST. | Up to 6 months
  An evaluable patient will be classified as a responder if the patient achieves a partial response (PR), complete response (CR) or stable disease (SD) ≥ 4 cycles.

SECONDARY OUTCOMES:
Progression free and overall survival | Progression-Free Survival (PFS) is defined as the duration of time from the start of treatment to the time of objective progression or death. [Time Frame: Up to 4 years]
  Determined using the Kaplan-Meier method with PFS at important time points reported along with 95% two sided confidence intervals.
Define and describe the toxicities of selumetinib in combination with sirolimus in patients with unresectable or metastatic NF1 associated or sporadic MPNST. | Up to 6 months
  This study will use CTEP Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 for toxicity and adverse event reporting. The toxicities will be graded and summarized descriptively and tabulations on the type, severity and relationship to study treatment will be performed.
Assess the impact on pain interference | Up to 6 months
  Pain interference metrics will be assessed using the Patient Reported Outcomes Measurements Information System (PROMIS) scale to assess the impact of pain on daily activities. This is a self-report measure that assesses the degree to which pain has interfered with the ability to complete daily activities over the past 7 days. Items are rated on a 5-point Likert scale and the measures yield standardized T-scores.
Assess the impact on pain severity | Up to 6 months
  Pain metrics will be assessed using the Numerical Rating Scale-11 (NRS-11) scale to assess pain severity. The scale consists of a horizontal line with 0 representing "no pain" and 10 representing "worst pain you can imagine." Patients will circle one number from 0 to 10 that best describes how much their tumor pain hurt during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute; Brigitte Widemann, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri